CLINICAL TRIAL: NCT03970980
Title: Increasing FIO2 Influences Accuracy of Fick-based Assessments of Cardiac Output in Cardiac Surgery Patients
Brief Title: FIO2 Influences Accuracy of Fick-based Cardiac Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201900558B0
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Output
Keywords: Fick Principle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIO2 >90% group (Experimental): This group receives FIO2 >90% during the surgery.
  Interventions: Other: fraction of inspired oxygen (FIO2)
- FIO2 <70% group (Active Comparator): This group receives FIO2 <70% during the surgery.
  Interventions: Other: fraction of inspired oxygen (FIO2)

INTERVENTIONS:
Other: fraction of inspired oxygen (FIO2) — Different group receives different (70% vs. 90%) fraction of inspired oxygen (FIO2) during the surgery.

SUMMARY:
Cardiac output (CO) monitoring is often required for clinical evaluation and management in critically ill patients and during anesthesia. There are many methods to measure CO. Fick-based CO estimation (Fick-CO) is one of the most commonly used methods, while thermodilution (TD-CO) is viewed as golden standard. But Fick-CO is still widely used, especially in catheterization laboratories and pediatric cardiologic department, whose patients often with congenital heart disease. Multiple studies from the 1960s find a strong correlation between TD-CO and Fick-CO. However, more recent studies reject the conclusion. Since Fick-CO is the ratio of oxygen consumption (V'O2) to the arteriovenous difference in oxygen content, many parameters are included in the Fick equation, such as V'O2, hemoglobin (Hb), arterial oxygen saturation (SaO2), mixed venous oxygen saturation (SvO2), partial pressure of arterial oxygen (PaO2), and mixed venous oxygen tension (PvO2). Any changes of each parameter may influence the accuracy of Fick-CO calculation. This may be the reason why it remains controversial whether Fick-CO and TD-CO are interchangeable or not. Although there are lots of studies comparing Fick-CO and TD-CO, discussing the impact of V'O2 on Fick-CO, how the other parameters influence the final CO estimation are rarely focused. Therefore, the purpose of this study was to assess the influence of FIO2 on PaO2, SvO2, PvO2, and the accuracy of Fick-CO in cardiac surgery patients.

DETAILED DESCRIPTION:
Patients who are aged ≥20 years, are undergoing planned elective cardiac surgery, and provided signed informed consent are included in the present study. Any patients with cardiac arrhythmia or an intra-cardiac shunt are excluded.

The patients are randomly assigned to 2 groups: FIO2 <70% or FIO2 >90%. And during the surgery, the oximeter values are kept ≥98%. Intra-operatively, FIO2, PaO2, SvO2, PvO2, Hb, and TD-CO are recorded.

ELIGIBILITY:
Inclusion Criteria:

* undergoing planned elective cardiac surgery
* agree to sign informed consent

Exclusion Criteria:

* cardiac arrhythmia
* intra-cardiac shunt

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
The Hemoglobin Values in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will collect hemoglobin data in each patient.
The Hemoglobin Values in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will collect hemoglobin data in each patient.
The Oxygen Consumption in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will calculate oxygen consumption in each patient.
The Oxygen Consumption in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will calculate oxygen consumption in each patient.
The SaO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record SaO2 data in each patient.
The SaO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record SaO2 data in each patient.
The SvO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record SvO2 data in each patient.
The SvO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record SvO2 data in each patient.
The PaO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record PaO2 data in each patient.
The PaO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record PaO2 data in each patient.
The PvO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record PvO2 data in each patient.
The PvO2 in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  The patients were divided into two FIO2 groups (FIO2 >90% or <70%) during the surgery. We will record PvO2 data in each patient.

SECONDARY OUTCOMES:
The Precision of Fick-based Cardiac Output in Different FIO2 Groups during Cardiac Surgeries | 5 minutes before surgical incision
  After collecting the elements data included in the Fick eqaution (oxygen consumption, hemoglobin, SaO2, SvO2, PaO2, and PvO2), we can calculate the Fick-based cardiac output in each patient. And the pulmonary artery thermodilution is adopted as the standard cardiac output monitoring method. We will calculate the correlation and level of agreement between Fick-based cardiac output and pulmonary artery thermodilution in the two groups.
The Precision of Fick-based Cardiac Output in Different FIO2 Groups during Cardiac Surgeries | 5 minutes after finishing protamine infusion
  After collecting the elements data included in the Fick eqaution (oxygen consumption, hemoglobin, SaO2, SvO2, PaO2, and PvO2), we can calculate the Fick-based cardiac output in each patient. And the pulmonary artery thermodilution is adopted as the standard cardiac output monitoring method. We will calculate the correlation and level of agreement between Fick-based cardiac output and pulmonary artery thermodilution in the two groups.

IPD SHARING:
Plan to Share IPD: Undecided